CLINICAL TRIAL: NCT00366990
Title: Clinical Trial to Reverse Early Arterial Stiffening
Brief Title: Low Sodium Diet and Behavioral Intervention for Reversing Arterial Stiffening in Overweight Individuals
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emma Barinas-Mitchell, PhD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 415; 5R01HL077525 (NIH)
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Obesity
Keywords: Arterial Stiffening
MeSH Terms: conditions — Cardiovascular Diseases; Obesity | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- weight loss and sodium intake reduction (Active Comparator): Behavioral and weight loss intervention, including a low sodium diet. Study goals are a 10% weight loss, 200 minutes of moderate physical activity a week, such as walking, and a 50% reduction in sodium intake.
  Interventions: Behavioral: Low Sodium Diet
- weight loss and normal sodium intake (Placebo Comparator): Behavioral and weight loss intervention, with regular sodium intake. Study goals are a 10% weight loss, 200 minutes of moderate physical activity a week, such as walking.
  Interventions: Behavioral: Regular Sodium Intake

INTERVENTIONS:
Behavioral: Low Sodium Diet — Group sessions once a week for 16 weeks, bi-weekly for 16 weeks, and monthly for 16 weeks on behavioral & weight loss topics with a focus on lowering sodium intake.
  Arms: weight loss and sodium intake reduction
Behavioral: Regular Sodium Intake — Group sessions once a week for 16 weeks, bi-weekly for 16 weeks, and monthly for 16 weeks on behavioral & weight loss topics.
  Arms: weight loss and normal sodium intake

SUMMARY:
Obese individuals are at risk for developing cardiovascular disease (CVD). Increasing physical activity, losing weight, and reducing sodium intake may reverse arterial stiffness and blood vessel damage that is linked to obesity. This study will evaluate the effectiveness of a low sodium diet and a behavioral weight loss intervention in reducing arterial stiffness in overweight young adults.

DETAILED DESCRIPTION:
CVD includes diseases that affect the heart and blood vessels. Arterial stiffness, in which arteries harden and become less flexible, increases the risk of developing CVD. Arterial stiffness increases both with age and in certain disease states, including high blood pressure, diabetes, and obesity. Young adults who are obese prematurely place themselves at risk for developing arterial stiffness and CVD. Physical activity and weight loss may reverse arterial stiffness in these individuals. Reducing sodium intake, which has been proven to decrease blood pressure, may also improve blood vessel function and arterial stiffness. The purpose of this study is to evaluate the effectiveness of a low sodium diet and a behavioral weight loss intervention in reducing arterial stiffness in young, moderately overweight individuals.

Participants will first attend a baseline study visit, at which time blood will be collected, and height, weight, waist circumference, and blood pressure will be measured. Questionnaires to assess medical history, physical activity levels, and dietary habits will be completed. An ultrasound will be used to evaluate blood vessel function and arterial stiffness. All participants will then take part in a 12-month behavioral and dietary intervention. The intervention will emphasize increasing physical activity and decreasing caloric intake by modifying lifestyle choices, physical and social environments, and attitudes toward food and exercise. Participants will be randomly assigned to follow either a low sodium diet or a normal sodium diet. During Months 1 through 4, participants will attend weekly study visits for group counseling sessions; during Months 4 through 8, study visits will occur once every two weeks; and during Months 8 through 12, they will occur once a month. At each study visit, weight, waist circumference, and blood pressure will also be measured. If necessary, individual counseling sessions will be scheduled. Participants will also document daily physical activity and caloric intake in a diary. Baseline evaluations will be repeated at Months 6, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 35

Exclusion Criteria:

* High blood pressure currently being treated with medication
* Blood pressure greater than or equal to 140/90 mm Hg on two consecutive study visits
* Diabetes, defined as either a fasting glucose test result of .126 or current use of hypoglycemic medications
* Currently taking hyperlipidemia medication
* Currently taking vasoactive medications
* History of known atherosclerotic disease (e.g., angina, heart attack, lower extremity arterial disease)
* Underlying inflammatory condition (e.g., systemic lupus erythematosus, rheumatoid arthritis)
* Chronic infection
* Current participation in a formal exercise or weight loss program
* Pregnant or planning to become pregnant during the study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 349 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | Measured at Month 6

SECONDARY OUTCOMES:
Arterial stiffness and remodelling | Measured at Months 6, 12 and 24
Endothelial function | Measured at Months 6, 12, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barinas-Mitchell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cooper JN, Tepper P, Barinas-Mitchell E, Woodard GA, Sutton-Tyrrell K. Serum aldosterone is associated with inflammation and aortic stiffness in normotensive overweight and obese young adults. Clin Exp Hypertens. 2012;34(1):63-70. doi: 10.3109/10641963.2011.618200. Epub 2011 Oct 18. PMID 22007645
- [Result] Cooper JN, Fried L, Tepper P, Barinas-Mitchell E, Conroy MB, Evans RW, Mori Brooks M, Woodard GA, Sutton-Tyrrell K. Changes in serum aldosterone are associated with changes in obesity-related factors in normotensive overweight and obese young adults. Hypertens Res. 2013 Oct;36(10):895-901. doi: 10.1038/hr.2013.45. Epub 2013 May 9. PMID 23657296
- [Result] Cooper JN, Evans RW, Mori Brooks M, Fried L, Holmes C, Barinas-Mitchell E, Sutton-Tyrrell K. Associations between arterial stiffness and platelet activation in normotensive overweight and obese young adults. Clin Exp Hypertens. 2014;36(3):115-22. doi: 10.3109/10641963.2013.789045. Epub 2013 May 8. PMID 23654212
- [Result] Cooper JN, Buchanich JM, Youk A, Brooks MM, Barinas-Mitchell E, Conroy MB, Sutton-Tyrrell K. Reductions in arterial stiffness with weight loss in overweight and obese young adults: potential mechanisms. Atherosclerosis. 2012 Aug;223(2):485-90. doi: 10.1016/j.atherosclerosis.2012.05.022. Epub 2012 May 30. PMID 22703865
- [Result] Njoroge JN, El Khoudary SR, Fried LF, Barinas-Mitchell E, Sutton-Tyrrell K. High urinary sodium is associated with increased carotid intima-media thickness in normotensive overweight and obese adults. Am J Hypertens. 2011 Jan;24(1):70-6. doi: 10.1038/ajh.2010.113. Epub 2010 May 27. PMID 20508622
- [Result] Lee JJ, Woodard GA, Gianaros PJ, Barinas-Mitchell E, Tepper PG, Conroy MB. Ectopic adiposity is associated with autonomic risk factors and subclinical cardiovascular disease in young adults. Obesity (Silver Spring). 2015 Oct;23(10):2030-6. doi: 10.1002/oby.21138. Epub 2015 Sep 3. PMID 26333626
- [Result] Hughes TM, Althouse AD, Niemczyk NA, Hawkins MS, Kuipers AL, Sutton-Tyrrell K. Effects of weight loss and insulin reduction on arterial stiffness in the SAVE trial. Cardiovasc Diabetol. 2012 Sep 22;11:114. doi: 10.1186/1475-2840-11-114. PMID 22998737
- [Result] Niemczyk NA, Catov JM, Barinas-Mitchell E, McClure CK, Roberts JM, Tepper PG, Sutton-Tyrrell K. Nulliparity is associated with less healthy markers of subclinical cardiovascular disease in young women with overweight and obesity. Obesity (Silver Spring). 2015 May;23(5):1085-91. doi: 10.1002/oby.21044. Epub 2015 Apr 10. PMID 25866258
- [Result] Hawkins M, Gabriel KP, Cooper J, Storti KL, Sutton-Tyrrell K, Kriska A. The impact of change in physical activity on change in arterial stiffness in overweight or obese sedentary young adults. Vasc Med. 2014 Aug;19(4):257-263. doi: 10.1177/1358863X14536630. Epub 2014 May 30. PMID 24879662
- [Result] Smith HA, Storti KL, Arena VC, Kriska AM, Gabriel KK, Sutton-Tyrrell K, Hames KC, Conroy MB. Associations between accelerometer-derived physical activity and regional adiposity in young men and women. Obesity (Silver Spring). 2013 Jun;21(6):1299-305. doi: 10.1002/oby.20308. PMID 23408709
- [Derived] Lott MP, Kriska A, Barinas-Mitchell E, Wang L, Storti K, Winger DG, Conroy MB. Impact of Lifestyle Strategies on Longer-Term Physical Activity and Weight. J Phys Act Health. 2017 Aug;14(8):606-611. doi: 10.1123/jpah.2016-0508. Epub 2017 Apr 19. PMID 28422536